CLINICAL TRIAL: NCT01938261
Title: The Preterm Infants' Paracetamol Study
Acronym: PreParaS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Outi Aikio, Specialist in Pediatrics and Neonatology, M.D., Ph.D., University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 100-2013; 2013-001842-33 (EudraCT Number)
Record Dates: First submitted 2013-08-22; First posted 2013-09-10 (Estimated); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Persistent Ductus Arteriosus; Complication of Prematurity; Pain or Discomfort in Intensive Care of Preterm Infants
MeSH Terms: conditions — Ductus Arteriosus, Patent; Pain | interventions — Acetaminophen; Saline Solution; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Paracetamol effect on ductus (Experimental): The first drug dose is given before 24 hours of age. Masked study drug is paracetamol infusion solution 10 mg/mL (PERFALGAN ®) or placebo, 0.45% saline solution. The loading dose is 20 mg/kg and the maintenance dose 7.5 mg kg every 6 hours for 4 days.
  Interventions: Drug: paracetamol; Drug: 0.45 % saline solution
- Paracetamol effect on pain (Experimental): The first drug dose is given before 24 hours of age. Masked study drug is paracetamol infusion solution 10 mg/mL (PERFALGAN ®) or placebo, 0.45% saline solution. The loading dose is 20 mg/kg and the maintenance dose 7.5 mg kg every 6 hours for 4 days.
  Interventions: Drug: paracetamol; Drug: 0.45 % saline solution

INTERVENTIONS:
Drug: paracetamol
  Other Names: Perfalgan 10 mg/ml infusion solution; Paracetamol Fresenius Kabi 10mg/ml
Drug: 0.45 % saline solution — Placebo
  Other Names: Natriumklorid Braun 4.5mg/ml solution

SUMMARY:
Present randomized, controlled, double-blind trial investigates the efficacy and safety of early (<24 h) intravenous paracetamol therapy for pain medication in very small premature infants. This phase 2 drug study focuses on the efficacy and safety of short-term use. The pharmacokinetics and pharmacodynamics of paracetamol, as well as the long-term effects, are studied.

This study recruits preterm infants born less than 32 weeks gestational age and treated at the neonatal intensive care unit of Oulu University Hospital. The informed consent is asked from all parents. The first drug dose is given before 24 hours of age. Masked study drug is paracetamol infusion solution 10 mg/mL or placebo, 0.45% saline solution. The loading dose is 20 mg/kg, and the maintenance dose 7.5 mg/kg every 6 hours for 4 days. The exact date of the closure of ductus is studied by repeated echocardiographic examinations. The symptoms of pain are screened by a pain scale of preterm infants (NIAPAS). Patients are monitored for signs of possible side effects. After discharge from hospital, patients are examined at follow-up clinic for the first year every 3 months and at 2 years of age.

DETAILED DESCRIPTION:
1 Hypotheses and aims: The aim of the present study is to evaluate the safety and efficacy of intravenous paracetamol in pain medication for small preterm infants in a randomized, controlled, double-blind trial. The primary outcome of the pain medication arm is the need for morphine medication (doses). The secondary outcomes are paracetamol serum concentrations, the side effects of paracetamol (possible hepatic dysfunction), neonatal and long-term morbidity, and mortality.

The primary outcome in the phase 2 ductus study-arm was diminishing of the ductal caliber at 5 days postnatal age. This study arm has been finalized and the results were published on 2016 (Härkin et al).

Hypotheses:

I. Hypothesis. Early, intravenous paracetamol is effective and safe therapy in the relief of pain and discomfort of a preterm infant.

II. Hypothesis. Paracetamol levels of a preterm infant remain in safety limits with study dosages.

III. Hypothesis. Early, intravenous paracetamol does not increase long-term morbidity in preterm infants.

Objectives:

1. Aim: to evaluate in a randomized, controlled, double-blind trial, the efficacy and safety of the early (<24 h), intravenous paracetamol in pain treatment of a preterm infant.
2. Aim: to evaluate the safety of the early (<24 h), intravenous paracetamol in preterm infants requiring intensive care.
3. Aim: to study pharmacokinetics and pharmacodynamics of paracetamol in a preterm infants
4. Aim: to evaluate the long-term effects of the early (<24 h), intravenous paracetamol in preterm infants requiring intensive care.

2 Study permissions: The research plan is registered to the investigational diary of the Department of Pediatrics, Oulu University Hospital (diary number 100-2013). For the present trial, the permissions from The Northern Ostrobothnia Hospital district's Ethical Board and Oulu University Hospital's administrative officials have been applied and granted. The study permission has been applied and granted from Fimea, the Finnish Medicines Agency. The amendment of the research plan was approved on 30.4.2018. This project has been assigned to EudraCT network (European Clinical Trials Database), Eudra CT number 2013-008142-33, and the international ClinicalTrials.gov registry, identification number NCT01938261.

Written informed consent is asked by the primary investigators of the study from all study patients' parents. The present clinical trial is managed by the principles of Good Clinical Practice, GCP (Fimea, act 2/2012, Clinical drug trials). The essential changes of the research plan are announced to Fimea according to the Drug legislation act 87a, using the European commission internet site (http://ec.europa.eu/health/documents/eudralex/vol-10/).

3 Sample size: The sample size calculation for the pain medication trial was checked after the first randomization. According to our previous study (Härmä et al, 2016), non-exposed premature infants received approximately 5 doses of morphine (SD 12) during their stay in the NICU. In order to treat infants without opioids, the clinical difference was approximated to be 6 doses. Therefore, with 20% power and 0.05 alpha-error, 126 infants (63/group) were required.

4 Study patients and exclusion criteria: This study will recruit all the intubated premature infants born less than 32 weeks of gestational age managed in Oulu University Hospital's neonatal intensive care unit. The deadline for recruitment and administration of the first dose of the study drug is postnatal age of 24 hours. The study exclusion criteria are severe structural, or chromosomal abnormality, and other severe clinical situation, which essentially affects the small premature infants' conventional early-stage treatment, e.g. severe asphyxia or persistent pulmonary hypertension (PPHN).

5 Randomization and blinding: As the informed consent is given, the study patient receives a trial number from the list made prior to the entry of the study. The trial number will match with an envelope where has been drawn a leaflet with the patient's study medication group written on it. Placebo, 0.45 % saline, is similar to paracetamol, both being clear liquids, so the staff will remain unaware which drug the patient receives. The study medication will be kept and prepared at the ward 55 in a separate office, in a locked cabinet. The study drug will be prepared by the study nurse, or by a nurse who does not participate in the study patients' treatment in any way.

6 Intervention: Masked study drug is 10 mg/ml paracetamol solution (Paracetamol Kabi Pharmacia®). Placebo is 0.45% saline solution, which does not enhance the potential small preterm infants' early-stage hypernatremia or hyperglycemia. Both are visually similar, clear solutions. Loading dose, 20 mg/kg, is followed by a maintenance dose 7.5 mg/kg every 6 hours, for four days. According to the earlier phase 1 studies, this dose is considered to be safe for small preterm infant. The drug is administered as a 15-minute infusion. No other paracetamol preparations are allowed to be given simultaneously with the study drug. After the intervention, the use of paracetamol should be restricted as far as it is possible. If the patient's clinical condition requires starting of paracetamol medication, there should be at least two days absence of paracetamol after the last dose of study medication. Half-life of intravenous paracetamol in neonates is about 4.5 hours. No other restrictions on the patient's therapy are set. After the study intervention, the patient is treated by the attending physicians' clinical judgment. Whenever necessary, the patient will be given the normal dose of morphine, 0.1 mg/kg.

6.1 Monitoring of the pain symptoms: The pain or discomfort of the patients will be screened using NIAPAS scoring before and after the study drug administration. According to the NIAPAS guidelines, values >5 indicate the need for evaluation for pain relief, either with using the non-medical pain relief methods, or increasing the pain medication dose. All the study patients will receive necessary pain medication during the study which would be morphine ad 0.1 mg/kg single doses, or morphine infusion. All morphine doses given during and after the intervention are recorded and calculated as the cumulative dosage.

7 Paracetamol safety: Using the study drug dosage, no signs of liver or renal failure have been described before. In addition, in the recent retrospective analysis among the study unit patient population, none of the preterm infants who received paracetamol showed any clinical or laboratory signs of either complication. No increased levels of liver transaminases, bilirubin or creatinine were detected.

In paracetamol intoxication, the hepatic failure is caused by a paracetamol metabolite, not paracetamol itself. Thus, the symptoms of intoxication are not immediately evident. The hepatic tissue damage can be prevented administering the paracetamol antidote as soon as possible. Even a suspicion of a possible intoxication in an otherwise symptom-free patient is to be taken seriously. This situation should be cautiously clarified, and, if necessary, the antidote started vigorously.

The signs and symptoms of paracetamol intoxication include:

* During the first 24 hours, nausea, vomiting, loss of appetite, fatigue, and perspiration may be manifested.
* 24-48 h after the overdose, the signs of it may be seen in the laboratory examinations: bilirubin and hepatic transaminase levels increase, and the prothrombin time lengthens (INR increases; this may happen without hepatic failure if the synthesis of vitamin K dependent coagulation factors is inhibited). Diuresis may be diminished due to possible dehydration (vomiting), renal failure, and the antidiuretic action of paracetamol.
* 2-5 days later, the liver and renal tissue damage develops. In the patients with hepatic failure, metabolic acidosis is usually seen.

Early acetyl cysteine therapy (<16 h after the overdose) may inhibit the hepatic failure, but even when started later, the tissue damage may be restricted. If necessary, the Poison Information Centre is consulted about the individualized instructions for treatment. The initial treatment includes intravenous fluid therapy in order to correct the acidosis, and the goal for the diuresis would be >1.5 ml/kg/h. The intravenously administered study medication cannot cause any harmful effects to the patients' relatives, the hospital staff, or the environment.

8 Monitoring, reporting and follow-up of the possible side effects: All study patients will be monitored for signs of possible side effects, especially the signs of hepatic or renal dysfunction. During the first postnatal days, serum bilirubin levels and diuresis will be followed. If a patient had prolonged or otherwise pronounced jaundice, the abdominal ultrasound would be performed. Any evidence of hepatic or renal dysfunction would be an indication to withdraw the study medication, and to measure the hepatic transaminases and creatinine concentrations. Symptomatic hepatic or renal failure is defined as an emergency when the blinding code could be opened and the study discontinued.

All harmful events and suspected side effects are individually evaluated for possible association to the study drug. The associations are classified: certain - likely - unlikely - not possible. The harmful events that are classified significant (SUSAR) are listed by the responsible investigator. Of the serious and unexpected harmful events, death or mortal danger are announced to Fimea within seven days after the incidence and the others within 15 days. The list of the harmful events is delivered to Fimea every year.

9 Pharmacokinetics: From those study patients with an arterial cannula, a single 1 ml blood sample at 48 hours postnatal age will be collected to evaluate paracetamol serum concentrations and the biological effects of prematurity. Of all the routine blood samples, any remaining droplets are retained for paracetamol concentration measurements.

10 Data collection: The study data will be collected using Centricity Critical Care Clinisoft software (GE Healthcare). All the data is confidential. All the study personnel are involved with confidentiality. The computed data is collected into the hospital's intranet station O. Study papers are mapped, and kept in the room of the responsible investigator. The Office of the Data Protection Ombudsman has been informed about the study register. The study results will be published in international, peer-reviewed medical literature, and in medical theses.

11 Quality control: An external study monitor, observing the quality of the methods used and the fulfillment of the study patients' rights, has been named.

12 Long-term follow-up: For the first year after discharge from hospital, the patients will be examined every three months at the follow-up clinic. Patients will be examined the clinical status, basic laboratory parameters, and if necessary, radiographic studies.

13 Statistical analyses: The intention-to-treat principle is applied in all analyzes. P-value <.05 will be considered significant. Statistical analyzes will be made using the IBM SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants born < 32 weeks gestational age

Exclusion Criteria:

* congenital malformation
* lethal disease
* chromosomal abnormality
* persistent pulmonary hypertension of a newborn

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2013-08 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Ductus diameter mm/kg | at postnatal age of 5 days
  Measured by cardiac ultrasound
Cumulative dosage of morphine | at postnatal age of 5 days
  The amount of morphine doses administerd during the study

SECONDARY OUTCOMES:
Number of patients who received any treatment for persistent ductus arteriosus | participants will be followed for the duration of NICU stay, an expected average of 12 weeks
  Prescribed by an attending clinician
Postnatal age of ductus closure | participants will be followed for the duration of NICU stay, an expected average of 12 weeks
  The date of the cardiac ultrasound examination when ductus was judged closed
Left atrium to aorta ratio | participants will be followed for the duration of NICU stay, an expected average of 12 weeks
  Measured by cardiac ultrasound
Number of apneic periods/day | up to 5 days postnatal age
  Apneas requiring stimulation by nurses
NIAPAS screening scores | up to 5 days postnatal age
  Scale 2-18, according to Polkki et al
Duration of mechanical ventilation | participants will be followed for the duration of NICU stay, an expected average of 12 weeks
  The number of days from intubation to extubation

OTHER OUTCOMES:
Long-term morbidity diagnoses | participants will be followed until 40 weeks gestational age, an expected average of 16 weeks
  BPD; ROP; ICH; NEC
Mortality | participants will be followed until 40 weeks gestational age, an expected average of 16 weeks
  Death cases
Paracetamol side effects | participants will be followed until 40 weeks gestational age, an expected average of 16 weeks
  Adverse reactions linked to IMP
Paracetamol serum concentrations | up to 5 days postanatal age
  Measured paracetamol serum levels

CONTACTS AND LOCATIONS:
Overall Officials: Timo Saarela, M.D., Ph. D., Principal Investigator — Oulu University Hospital; Mikko Hallman, M.D., Ph.D., Study Chair — University of Oulu
Locations (1):
- Department of Pediatrics, Oulu University Hospital, Oulu, Finland

REFERENCES:
- [Derived] Jasani B, Mitra S, Shah PS. Paracetamol (acetaminophen) for patent ductus arteriosus in preterm or low birth weight infants. Cochrane Database Syst Rev. 2022 Dec 15;12(12):CD010061. doi: 10.1002/14651858.CD010061.pub5. PMID 36519620
- [Derived] Harkin P, Harma A, Aikio O, Valkama M, Leskinen M, Saarela T, Hallman M. Paracetamol Accelerates Closure of the Ductus Arteriosus after Premature Birth: A Randomized Trial. J Pediatr. 2016 Oct;177:72-77.e2. doi: 10.1016/j.jpeds.2016.04.066. Epub 2016 May 20. PMID 27215779